CLINICAL TRIAL: NCT00217815
Title: A Phase Ib, Pharmacokinetic, Multiple Center, Open Label Study Evaluating the Safety and Efficacy of Mycograb Administered IV in Combination With Docetaxel in Metastatic or Recurrent Breast Cancer Patients
Brief Title: Preliminary Study of Mycograb and Docetaxel in Advanced Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NeuTec Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTP/ONC/001
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — efungumab; Docetaxel

INTERVENTIONS:
Drug: Mycograb, Docetaxel

SUMMARY:
The study hypothesis is that the addition of Mycograb to docetaxel will improve outcome in advanced carcinoma of the breast.

DETAILED DESCRIPTION:
Combination therapies that incorporate new agents have demonstrated the potential to improve outcome for patients with metastatic breast carcinoma. Docetaxel has been shown to be a very active drug in breast cancer, and anthracycline-based chemotherapy combinations represent the most active form of therapy generating objective response rates of between 40-70%. Mycograb® was most effective in breast carcinoma cell lines in combination with cisplatin, docetaxel and anthracyclines (doxorubicin, daunorubicin).

We propose that Mycograb® binds to hsp90, inhibiting hsp90 chaperone functioning and resulting in the destabilization of key proteins including estrogen/steroid receptors, nitric oxide synthase, ras1, MAP (Mitogen-activated protein) kinase, Src, Erb-B2,(erythroblastic leukemia viral oncogene homolog 2) HER(human estrogen receptor) kinases and EGFR (epidermal grown factor receptor). Over expression of HER2 receptors are observed in malignancies such as breast cancer and reportedly have been associated with resistance to chemotherapeutic agents. Both maturing and fully mature forms of the receptor depend on hsp90 association for stability. Inhibition of hsp90 function down regulates AKT kinase and Src kinase which are non-receptor kinase. Therefore, Mycograb® may be of use in estrogen dependent and hormone independent breast cancers.

Mycograb® has been demonstrated to have anti-tumor activity in cell culture. The 50% cytotoxicity of Mycograb® on its own is 50 Combination therapies that incorporate new agents have demonstrated the potential to improve outcome for patients with metastatic breast carcinoma. Docetaxel has been shown to be a very active drug in breast cancer, and anthracycline-based chemotherapy combinations represent the most active form of therapy generating objective response rates of between 40-70%. Mycograb® was most effective in breast carcinoma cell lines in combination with cisplatin, docetaxel and anthracyclines (doxorubicin, daunorubicin).

We propose that Mycograb® binds to hsp90, inhibiting hsp90 chaperone functioning and resulting in the destabilization of key proteins including estrogen/steroid receptors, nitric oxide synthase, ras1, MAP kinase, Src, Erb-B2, HER kinases and EGFR. Overexpression of HER2 receptors are observed in malignancies such as breast cancer and reportedly have been associated with resistance to chemotherapeutic agents. Both maturing and fully mature forms of the receptor depend on hsp90 association for stability. Inhibition of hsp90 function down regulates AKT kinase and Src kinase which are non-receptor kinase. Therefore, Mycograb® may be of use in estrogen dependent and hormone independent breast cancers.

Mycograb® has been demonstrated to have anti-tumor activity in cell culture. The 50% cytotoxicity of Mycograb® on its own is 50 µg/ml (MCF7 [Breast cancer cell line designation]). Mycograb® in combination with docetaxel, doxorubicin and cisplatin and Herceptin increased the cytotoxicity in breast cancer cells.

It is appropriate to evaluate the apparent tumor response and survivor benefits resulting from the addition of Mycograb® to a docetaxel containing chemotherapy regimen in metastatic or recurrent breast cancer patients.

(MCF7). Mycograb® in combination with docetaxel, doxorubicin and cisplatin and Herceptin increased the cytotoxicity in breast cancer cells.

It is appropriate to evaluate the apparent tumor response and survivor benefits resulting from the addition of Mycograb® to a docetaxel containing chemotherapy regimen in metastatic or recurrent breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be female between the ages of 18 to 70 years old.
2. Patients must have histologically or clinically confirmed metastatic and/or recurrent breast cancer amenable to treatment with docetaxel.
3. Patients must have presence of at least one uni-dimensional measurable lesion with minimal lesion size > 20 mm at the largest diameter.
4. Patients may have had one previous chemotherapy regimen and must not have received prior chemotherapy with docetaxel.
5. Patients must have been off all hormonal therapy for at least 2 weeks prior to initiation of therapy.
6. Patients must have been off all chemotherapy or radiotherapy regimens for at least 4 weeks prior to initiation of chemotherapy.
7. Patients must have a life expectancy of at least 6 months.
8. Patients must have a ECOG status of 0, 1 or 2.
9. Patients must be willing to complete all procedures and visits as outlined in the protocol.
10. Patients must sign an informed consent form.
11. Patients must have negative blood test for HIV and hepatitis B and C.
12. Female patients of child bearing potential should use an effective method of contraception.

Exclusion Criteria:

1. Patients with brain or meningeal metastases.
2. Patients whose only measurable lesion is in the bone.
3. Patients with clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, respiratory, neurologic, psychiatric, immunologic, gastrointestinal, hematologic, metabolic or any other condition or laboratory abnormality that in the opinion of the investigator makes the patient unsuitable for participation in the study.
4. Patients with history of seizure disorder.
5. Patients who have received treatment with any other investigational drug within the preceding one month.
6. Patients who are pregnant or breast feeding.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-09; Study Completion 2006-10

PRIMARY OUTCOMES:
Impact on tumour size when compared to historical controls

SECONDARY OUTCOMES:
Safety data
Pharmacokinetics data

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pluzanska, MD, Principal Investigator — University of Lodz
Locations (3):
- Chemotherapie Clinic of Medical University Lodz, Lodz, Pabianicka, Poland
- Serbia (2):
  - Clinical Hospital Centre Bezanijska Kosa, Bezanijska Kosa Bb, Belgrade
  - Institute For Oncology and Radiology of Serbia, Pasterova 14, Belgrade